CLINICAL TRIAL: NCT06317532
Title: Effect of Functional Exercises on Pain and Quality of Life in Females With Primary Dysmenorrhea
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Manar Essam Al-Emary, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004766
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Primary Dysmenorrhea
Keywords: Primary Dysmenorrhea; Functional Exercises; Pain; Quality of Life
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle modification advice (Active Comparator): It will include 29 females suffering from primary dysmenorrhea. They will be asked to follow lifestyle modification advice during the program duration.
  Interventions: Other: Lifestyle modification advice
- Lifestyle modification advice + Functional exercises (Experimental): It will include 29 females suffering from primary dysmenorrhea. They will be given the same lifestyle modification advice as group A, in addition to performing a combination of various functional exercises (including two stretching exercises, one yoga position, two core-strengthening exercises, two pelvic area exercises, and Kegel exercises), for 45 minutes per session, three times /week for eight weeks.
  Interventions: Other: Lifestyle modification advice; Other: Functional exercises

INTERVENTIONS:
Other: Lifestyle modification advice — All female participants in groups A and B will be provided with lifestyle modification advice, including recommendations such as reducing caffeine intake, limiting salt consumption, decreasing animal fat consumption, quitting smoking, practicing relaxation techniques, applying heat when needed, considering the use of herbal agents, avoiding cold drinks and foods, and opting for loose, cotton clothing.
Other: Functional exercises — Each female in group (B) will perform the exercise program three times a week for eight weeks at the University Women's Health Unit Exercise protocols mainly consist of relaxation, strengthening, stretching, aerobic exercises, pelvic floor muscle strengthening exercises, yoga, and Pilates
  Arms: Lifestyle modification advice + Functional exercises

SUMMARY:
The aim of the study will be to investigate the effect of functional exercises on pain and quality of life in females with primary dysmenorrhea.

DETAILED DESCRIPTION:
Primary dysmenorrhea and menstrual pain are significant health, social and economic problems. It involves a broad spectrum of physical and emotional manifestations, with 50% to 91 % prevalence in young women.

Women with primary dysmenorrhea report significantly lower quality of life because of bodily pain, general health condition, and physical and social functioning. It compromises the most common gynecological alternations and is the primary cause of women's academic and work absenteeism, which reduces the quality of life, daily activities, and economic situation due to decreased working hours.

Non-Steroidal Anti-Inflammatory Drugs are the first therapeutic line for primary dysmenorrhea; however, they might be accompanied by undesirable side effects, such as dyspepsia, headache, and drowsiness.

So, there is a need for safe interventions with no side effects. Therefore, this study aims to investigate the effects of functional exercises on pain and quality of life in females with primary dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

1. Their ages will be ranged from 18 to 25 years
2. They will be suffering from primary dysmenorrhea based on the Menstrual Distress questionnaire.
3. Their BMI will be ranged from 20 to 25 kg/m2.
4. Having regular menstrual cycles (one every 28-34 days).
5. They will be sedentary virgin females.
6. They are non-smokers.
7. They have not been in any exercise program for three months.

Exclusion Criteria:

1. Having secondary dysmenorrhea.
2. Using regular medication or contraceptive pills.
3. Having neuromuscular, metabolic, or cardiac diseases.
4. Having a preexisting condition prevents them from engaging in an exercise program.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 58 (Estimated)
Dates: Start 2024-03-20 (Estimated); Primary Completion 2024-05-20 (Estimated); Study Completion 2024-05-20 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | 8 weeks
  It will be used to measure pain intensity for each female in both groups (A&B) before and after the end of treatment. The VAS is usually presented as a 10 cm horizontal line on which the participants' pain intensity is represented by a point between the extremes of "no pain at all "and "worst pain imaginable. " Its simplicity, reliability, and validity, as well as its ratio scale properties, make the VAS the optional tool for describing pain intensity.
The Menstrual Distress Questionnaire | 8 weeks
  It will be used to evaluate menstruation symptoms and distress for each female in both groups (A&B) before and after the end of treatment. It consists of symptoms or feelings associated with menstruation. The total number of items is 47. It is a 5-point rating scale from 0-4. Each item has five options, i.e., No, mild, moderate, severe, and very severe. An option of (very severe) has a score of 4, (severe) has a score of 3, (moderate) has a score of 2, (mild) has a score of 1, (No) has a score of 0. It includes seven subscales as (pain, water retention, autonomic reactions, negative affect, impaired concentration, mood and behavioral changes, and arousal control). The overall score was interpreted as follows: <50 - mild, 50 to 70 - moderate, and >70 severe.

SECONDARY OUTCOMES:
Quality of life enjoyment and satisfaction questionnaire | 8 weeks
  It will be used to assess health-related quality of life for participants of both groups (A&B) before and after the end of the treatment program. It consists of items that evaluate overall enjoyment and satisfaction regarding; Physical Health, mood, work, household and leisure activities, family and social relationships, ability to function in daily life, economic status, living or housing situation, ability to get around physically, ability to do work or hobbies, and overall sense of being. Responses will be scored on a five-point scale (from "very poor" to "very good"), where higher scores indicate better enjoyment and satisfaction with life. Scores will be added and presented as a percentage of the total maximum score. A percentage of the total score of > 70 represents the normal quality of life.
Pressure pain threshold assessment | 8 weeks
  A pressure algometry will be used to measure pressure pain thresholds for all participants in both groups (A&B) before and after the end of the treatment program.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Egypt